CLINICAL TRIAL: NCT03270293
Title: Efficacy and Tolerance Evaluation of a Bio-revitalizing Product Containing Hyaluronic Acid With High and Low Molecular Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1214
Record Dates: First submitted 2016-01-15; First posted 2017-09-01 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2016-01

CONDITIONS: Malar and Sub-malar Volume Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Profhilo (Experimental): The intradermal procedure was performed bilaterally on the face, at level of the following five points:
  1. zygomatic protuberance
  2. nostril's angle
  3. inferior margin of tragus
  4. lip marionette lines
  5. mandibular angle. The amount of product injected, was 0.2 ml for each injection-point.
  Interventions: Device: Profhilo

INTERVENTIONS:
Device: Profhilo
  Other Names: IBSA

SUMMARY:
Primary end point of the study was to evaluate clinically and by non-invasive instrumental evaluations tolerance and efficacy of a bio-revitalizing product containing hyaluronic acid with high (H-HA) and low (L-HA) molecular weight; the micro-injection of the study product was performed by a specialized dermatologist, bilaterally on the face (zygomatic protuberance, nostril's angle, inferior margin of tragus, lip marionette lines, mandibular angle) of healthy female volunteers aged 30-60 years.

It was also aim of this study to evaluate efficacy by the volunteers and tolerance both by investigator and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* age 30-60 years
* agreeing to present at each study visit without make-up
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study, without appropriate sun protection
* accepting to sign the Informed consent form.

Exclusion Criteria:

* pregnancy
* lactation
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study
* subjects not in menopause who do not accept to perform the pregnancy test during the basal visit, 4 and 8 weeks after the first biomineralising treatment execution
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 12 months prior to the study start
* performing permanent filler in the past
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test
* sensitivity to the test product or its ingredients (an accurate anamnestic assessment will performed by the investigator)
* subjects whose insufficient adhesion to the study protocol is foreseeable
* participation in a similar study actually or during the previous 3 months.
* presence of cutaneous disease on the tested area, as lesions, scars, malformations
* recurrent facial/labial herpes
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy.
* anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago)
* assumption of drugs able to influence the test results in the investigator opinion.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) improvement | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  Grade 1 (absent): no visible nasolabial fold; continuous skin line. Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.
Facial Volume Loss Scale (FVLS) improvement | 16 weeks
  Reduction of face volume loss corresponding to a decrease from the baseline of the Facial Volume Loss Scale (FVLS) where Grade 1 Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). No prominent bony landmarks. No visibility of underlying musculature.
  Grade 2 An intermediate point between grade 1 and grade 3. Grade 3 Moderate concavity of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas. Prominence of bony landmarks. May have visibility of underlying musculature.
  Grade 4 An intermediate point between grade 3 and grade 5. Grade 5 Severe indentation of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). Severe prominence of bony landmarks. Clear visibility of underlying musculature.
Surface microrelief's regularity improvement | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Improvement of skin surface microrelief corresponding to a reduction of the clinical score of microrelief's regularity grade where Grade 1:very regular, Grade 2: regular, Grade 3: irregular, Grade 4: very irregular.
  Clinical evaluation of surface microrelief's regularity grade is carried out on the digital picture acquired by FotoFinderDermoscope with a magnification of 20X
Determination of profilometric parameters | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Reduction of the nasolabial fold and marionette lines profilometric parameters versus baseline where Ra is average roughness of the analysed profile, Rt is wrinkles total high, Rv is wrinkles maximum depth.
  Replicas of nasolabial fold and marionette lines are obtained using silicone rubber. A picture of the skin replicas is taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to elaborate 3D representations of skin wrinkles as well as to measure skin principal profilometric parameters.
Skin plastoelasticity improvement | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Improvement of the principal torsiometric parameters Ue (immediate extensibility), Uf (final extensibility), Uv (viscoelasticity) and Ur (immediate elastic recovery).Skin firmness is measured with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK).
Superficial skin hydration improvement | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Improvement of skin electrical capacitance value measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany).
  The measure of the skin capacitance properties is an indirect expression of its hydration level.
Deep skin hydration improvement | Basal visit (T0), Week 4 (T4W) , Week 8 (T8W), Week 12 (T12W), Week 16 (T16W).
  Improvement of tissue dielectric constant value of superficial and deep skin layers measured with MoistureMeterD (Delfin Technologies, Kuopio - Finland)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL
Locations (1):
- DERMING, Monza, Monza-brianza, Italy